CLINICAL TRIAL: NCT06451536
Title: Prognostic Significance of Ga-68 FAPI PET Before Immunotherapy in Pleural Mesothelioma
Brief Title: Ga-68 FAPI PET Before Immunotherapy
Acronym: FAPBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Liv Hospital Ankara (Other); Social Sciences University of Ankara (Other); Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Cigdem Soydal, AsC Prof of Nuclear Medicine, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPBI Trial
Record Dates: First submitted 2024-05-17; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Mesotheliomas Pleural
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Intervention Model Description: prediction of immunotherapy response with Ga-68 FAPI PET
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients underwent Ga68 FAPI PET before immunotherapy
  Interventions: Diagnostic Test: Ga-68 FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: Ga-68 FAPI PET/CT — imaging of FAP expression of tumor before immunotherapy

SUMMARY:
It is aimed to evaluate FAP expression and its success in predicting treatment response before immunotherapy used in the treatment of malignant mesothelioma with Ga68 FAPI PET/CT imaging, which allows in vivo evaluation of FAP expression, which is thought to be associated with immunosuppression and resistance to immunotherapy.

DETAILED DESCRIPTION:
Patients diagnosed with pleural mesothelioma and planned for immunotherapy will be included in the study. Patients will undergo Ga68 FAPI PET/CT imaging within 10 days before the start of immunotherapy treatment, and SUVmax, SUVmean, metabolic tumor volume and total Ga68 FAPI uptake parameters will be obtained from the tumors. Following this, the routine treatment and follow-up of the patients will be carried out by their clinicians. It will be evaluated whether there is a correlation between treatment response and initial Ga-68 FAPI PET findings.

ELIGIBILITY:
Inclusion Criteria:

* Having a histopathologically confirmed diagnosis of
* Pleural Mesolthelioma
* Patients scheduled for immunotherapy with anti-PDL-1 and/or anti-CTLA-4 antibodies as first or second line therapy
* Patients who gave informed consent form to participate in the study

Exclusion Criteria:

* ECOG>2
* Patients who did not provide informed consent form to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Prediction of immune therapy response with Ga-68 FAPI PET | 6. month after initiation of therapy
  prediction of immunotherapy response with SUVmax measured with Ga-68 FAPI PET before immunotherapy
Prediction of immune therapy response with Ga-68 FAPI PET | 6. month after initiation of therapy
  prediction of immunotherapy response with total FAPI volume measured with Ga-68 FAPI PET before immunotherapy
Prediction of immune therapy response with Ga-68 FAPI PET | 6. month after initiation of therapy
  prediction of immunotherapy response with total lesion FAPI uptake measured with Ga-68 FAPI PET before immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)